CLINICAL TRIAL: NCT01586429
Title: Ultrasound Guided Femoral Nerve Block Catheter Analgesia Compared With Epidural Analgesia for Patients With Knee OA (Osteoarthritis) Who Underwent Unilateral Total Knee Replacement
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Dr. Tariq Alzahrani, Associate Professor, King Saud University
Other Study IDs: E-12-589
Record Dates: First submitted 2012-04-25; First posted 2012-04-26 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2011-02

CONDITIONS: Knee Osteoarthritis
Keywords: comparing the analgesic efficacy of ultrasound-guided nerve block catheter compared with epidural analgesia
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Analgesia, Epidural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Epidural
  Interventions: Other: Ultrasound guided femoral nerve block catheter analgesia compared with epidural analgesia for patients with knee OA (osteoarthritis)
- Femoral catheter
  Interventions: Other: Ultrasound guided femoral nerve block catheter analgesia compared with epidural analgesia for patients with knee OA (osteoarthritis)

INTERVENTIONS:
Other: Ultrasound guided femoral nerve block catheter analgesia compared with epidural analgesia for patients with knee OA (osteoarthritis)

SUMMARY:
Post-operative pain following total knee replacement can be disabling and sometimes lead to the need for prolonged hospital stay. Therefore development of improved post-operative modalities for total knee replacement surgery pain control is important. High-resolution ultrasound (US) allows accurate visualization of nerves and surrounding structures and can lead to higher success rates of nerve block. The investigators aim at comparing the analgesic efficacy of ultrasound-guided nerve block catheter compared with epidural analgesia for patients with knee OA who underwent unilateral total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

* Male / female, Bilateral or unilateral knee OA (Osteoarthritis), and ASA (American Society of Anesthesiologist classification) 1 and 2.

Exclusion Criteria:

* Bilateral total knee replacement, Revision total knee replacement, previous knee surgery, Rheumatoid Arthritis, Avascular necrosis (AVN) knee, Post traumatic or post infectious OA, ASA3 and 4.

Min Age: 30 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: for patients with knee OA (osteoarthritis) who underwent unilateral total knee replacement.
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Locations (2):
- Saudi Arabia (2):
  - King Saud University, Riyadh, Riyadh Region
  - King Saud University, Riyadh Region, Riyadh Region